CLINICAL TRIAL: NCT07051668
Title: The Right Call: Implementing a Sepsis Diagnostic Safety Toolkit in a Pediatric Transfer Call Center to Improve Diagnosis of Children in General Emergency Settings
Brief Title: The RightCall: Implementing a Sepsis Diagnostic Toolkit to Improve Pediatric Diagnosis in ED Transfer Calls
Acronym: RightCall
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-2340; 1R18HS029786-01 (AHRQ)
Record Dates: First submitted 2025-06-24; First posted 2025-07-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Diagnosis; Emergencies
Keywords: Pediatric, Diagnosis
MeSH Terms: conditions — Sepsis; Disease; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation Phase (usual care) (No Intervention): Historic standards of care were used by all clinicians during the 24-month pre-implementation phase. This can also be referred to as usual care.
- Post-implementation Phase (using Diagnostic Toolkit) (Active Comparator): The Pediatric Sepsis Diagnostic Toolkit will be used during the post-implementation phase to better diagnose sepsis in transfer cases.
  Interventions: Other: Pediatric Sepsis Diagnostic Toolkit

INTERVENTIONS:
Other: Pediatric Sepsis Diagnostic Toolkit — The toolkit consists of the following items: 1) a recommendation to request and report vital signs in all pediatric hospital/ED transfers, 2) dissemination of evidence based pediatric sepsis diagnostic criteria to accepting and referring providers and transfer nurses, and 3) accepting physician education in conversational strategies to promote improved diagnostic accuracy during pediatric transfer conversations.
  Arms: Post-implementation Phase (using Diagnostic Toolkit)

SUMMARY:
Sepsis is a leading cause of death in children, and an early diagnosis that improves outcomes is less likely in children who are treated in general Emergency Departments (EDs), that treat adults and children, compared to pediatric Emergency Departments. The study team, in collaboration with invested clinicians and expert partners, has developed a pediatric sepsis diagnostic safety toolkit that we will implement in a pediatric health system's transfer call center. Preparation for launch of the toolkit will include education throughout Children's Hospital Colorado (CHCO), with a focus on transfer center nurses and accepting CHCO physicians who will be partnering in delivering the toolkit. Usual avenues for clinical education will be used, including meetings, endorsement from clinical leaders, emails, and physical materials such as badge and pocket cards. Referring Emergency Department (ED) providers outside of CHCO will not receive education about the toolkit by design, since they are the recipients of the toolkit which is designed to disseminate sepsis diagnostic knowledge in real time to general EDs within existing transfer workflows. This research will test whether the toolkit improves early pediatric sepsis diagnosis in general EDs where most children receive their first critical hours of care.

DETAILED DESCRIPTION:
This study is a prospective type 2 hybrid implementation-effectiveness trial to evaluate a sepsis diagnostic safety toolkit. The study team will use explanatory mixed methods to assess quantitative and qualitative metrics, including PRISM contextual factors and RE-AIM outcomes such as accuracy, adoption, adaptations, sustainability, and context.

The study team will conduct a pre/post-evaluation of the toolkit to measure effectiveness outcomes; and also will evaluate additional implementation outcomes using quantitative and qualitative approaches.

The study will consist of a 24 month pre-intervention period and a 24-month post-intervention period, capturing the same sepsis seasonality during both phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients transferred to Children's Hospital Colorado (CHCO) for emergency or inpatient care, as identified in the extant CHCO transfer center database AND in the extant CHCO quality improvement sepsis database AND one of the following:
* Patients who met Phoenix sepsis criteria 1) in the referring ED, 2) during transport, 3) in the first 6 hours after arrival at the pediatric hospital, or 4) patients who developed Phoenix sepsis within 24 hours of arrival at the Children's Hospital underwent independent physician review by three emergency physicians. Patients in whom all three physicians agreed sepsis was most likely present, using the structured SaferDx tool were included

Exclusion Criteria:

* Patients less than one month of age
* Patients whose transfer call recording was not available in the database

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | measured at the end of the 24 month post-implementation period
  Proportion of included patients in whom all 3 of the following occur while the patient is physically in the referring hospital: 1) verbal or written use of the term "sepsis", 2) Intravenous antibiotics ordered,and 3) intravenous flue bolus ordered.

SECONDARY OUTCOMES:
Vital Signs Reported on Transfer Phone Call | measured at the end of the 24 month post-implementation period
  Proportion of included patients with any vital sign reported during the transfer phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Halden F. Scott, MD, MSCS, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient Electronic Health Record (EHR) data will be stored in Excel (csv) files for data analysis at University of Colorado. Cleaned and deidentified datasets in SAS or R statistical software will be shared upon request.
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT07051668/SAP_001.pdf